CLINICAL TRIAL: NCT02518308
Title: Mindfulness-Based Interventions in Patients Treated for Gynecologic Cancer - Impact on Patient Reported Outcomes and Immunologic Correlates
Brief Title: Mindfulness Intervention in Reducing Anxiety in Patients Who Have Been Treated for Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW15000; 2015-0549 (Other: Institutional Review Board); A532820 (Other: UW Madison); SMPH\OBSTET & GYNECOL\OB-GYN (Other: UW Madison); NCI-2015-01263 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-07

CONDITIONS: Anxiety; Cancer Survivor; Cognitive Impairment; Depression; Distress; Fatigue; Malignant Female Reproductive System Neoplasm; Pain; Sexual Dysfunction
MeSH Terms: conditions — Anxiety Disorders; Cognitive Dysfunction; Depression; Fatigue; Pain; Sexual Dysfunction, Physiological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Care Provider

ARMS (2):
- Arm I (MBSR intervention) (Experimental): Patients undergo an 8-week MBSR course, comprising weekly 2.5 hour classes and one 6-hour Saturday class at week 6 or 7. The MBSR program involves instruction in mindfulness meditation and yoga, and gives homework assignments involving practicing the well-being techniques taught in class. Patients are required to record and report time spent on home practice in a journal daily, and receive a weekly reminder to report their home practice.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Arm II (control) (No Intervention): Patients do not participate in the intervention, but are given the option to be placed on a waitlist for the MBSR course and may complete it within 6 months after the final study visit.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The Mindfulness-Based Stress Reduction program involves instruction in mindfulness meditation and yoga.
  Other Names: MBSR
  Arms: Arm I (MBSR intervention)

SUMMARY:
This pilot clinical trial studies how well a mindfulness-based stress reduction (MBSR) intervention works in reducing anxiety in patients who have undergone treatment for gynecologic cancer but no longer have any sign of disease. Gynecologic cancer is cancer of the female reproductive tract, which includes the cervix, endometrium, fallopian tubes, ovaries, uterus, and vagina. Side effects from treatment for these cancers may include anxiety, fatigue, depression, and sexual function changes. Mindfulness training uses meditation and yoga to help patients focus on breathing, bodily sensations, and mental awareness. This may help decrease patients' stress and anxiety and improve their quality of life, and may also help their immune system.

DETAILED DESCRIPTION:
Patients are randomized to 1 of 2 Arms.

ARM I (INTERVENTION): Patients undergo an 8-week MBSR course, comprising weekly 2.5 hour classes and one 6-hour Saturday class at week 6 or 7. The MBSR program involves instruction in mindfulness meditation and yoga, and gives homework assignments involving practicing the well-being techniques taught in class. Patients are required to record and report time spent on home practice in a journal daily, and receive a weekly reminder to report their home practice.

ARM II (WAIT-LIST CONTROL): Patients do not participate in the intervention, but are given the option to be placed on a waitlist for the MBSR course and may complete it within 6 months after the final study visit.

After completion of study, patients are followed up at 8 weeks (at completion of study) and 5 months (3 months from study completion).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any invasive gynecologic cancer without evidence of disease.
* Gynecologic cancer treatment (e.g., surgery, chemotherapy, radiation therapy) was completed within 5 years prior to date of enrollment.
* Able to speak, read and write English
* ECOG Performance Status between 0 and 3
* Subjects must have a phone.
* Experiencing 2 or more of the following symptoms felt to be associated (per the patient) with gynecologic cancer or previous gynecologic cancer treatment: anxiety (worry or feeling stressed), cognitive impairment (difficulty concentrating, focusing, memory loss), depression, existential/spiritual distress (hopelessness, lack of meaning in life, lack of peace), fatigue, pain, and sexual dysfunction. These symptoms may be new or worsened since cancer diagnosis. Both symptoms fomr this list must have been present one week prior to eligibility assessment, with worst severity rating greater than or equal to 3 (0-10 scale) for at least 1 of the 2 symptoms
* Expected to continue cancer care at UWCCC for the duration of the study.

Exclusion Criteria:

* Undergone cancer treatment (excluding hormonal therapy or biological maintenance therapy) in the 4 weeks prior to enrollment
* Expected to require cancer treatment, other than biologic or hormonal maintenance therapy, during the course of the study
* Any other cancer present within the last 5 years (other than gynecologic cancer under study and non-melanoma skin cancer)
* Practicing mindfulness meditation for an average of more than 1 hour/week or have taken mindfulness training in the past
* Documented history of Alzheimer's disease, dementia, or other neurologic deficit that could impact decision-making
* Prisoner or incarcerated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | Baseline to up to 5 months
  Measured by the 8-item anxiety subscale of the PROMIS scale.

SECONDARY OUTCOMES:
Change in depression | Baseline to up to 5 months
  Measured by PROMIS subscale for depression.
Change in fatigue | Baseline to up to 5 months
  Measured by PROMIS subscale for fatigue.
Change in sleep disturbance | Baseline to up to 5 months
  Measured by PROMIS subscale for sleep disturbance.
Change in sexual function | Baseline to up to 5 months
  Measured by Female Sexual Function Profile and Global Satisfaction with Sex Life questionnaire.
Change in existential/spiritual distress | Baseline to up to 5 months
  measured by Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being Scale (FACIT-SP-12 version 4)
Change in cognitive function | Baseline to up to 5 months
  Measured by the NIH Toolbox Assessments
Change in cortisol levels | Baseline to up to 5 months
  The biobehavioral link between MBSR intervention-related Quality of Life changes and immune cell function will be explored.
Change in levels of pro-inflammatory cytokines | Baseline to up to 5 months
  The biobehavioral link between MBSR intervention-related Quality of Life changes and immune cell function will be explored.
Change in immune cell phenotypes | Baseline to up to 5 months
  The biobehavioral link between MBSR intervention-related Quality of Life changes and immune cell function will be explored.
Change in NK cell function | Baseline to up to 5 months
  The biobehavioral link between MBSR intervention-related Quality of Life changes and immune cell function will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Spencer, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center Home Page — http://www.uwhealth.org/uw-carbone-cancer-center/cancer/10252